CLINICAL TRIAL: NCT05753696
Title: The Effect of Azilsartan in Patients With Diabetic Kidney Disease and Hypertension
Brief Title: Azilsartan in Patients With Diabetic Kidney Disease and Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-106
Record Dates: First submitted 2023-02-03; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Proteinuria; Kidney Dysfunction; Blood Pressure; Diabetic Kidney Disease
Keywords: diabetic kidney disease; hypertension
MeSH Terms: conditions — Proteinuria; Diabetic Nephropathies; Hypertension | interventions — azilsartan; Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- azilsartan group (Experimental): the initial dose of azilsartan is 20mg/day, if not reached the goal of blood pressure, azilsartan was adjust to 40mg/day
  Interventions: Drug: Azilsartan
- losartan group (Active Comparator): the initial dose of losartan is 40mg/day, if not reached the goal of blood pressure, losartan was adjust to 80mg/day
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan initial dose 20mg/d, if not reached the goal of hypertension; azilsartan dose 40mg/d
  Arms: azilsartan group
Drug: Losartan — losartan initial dose 40mg/d, if not reached the goal of hypertension; losartan 100mg/d
  Arms: losartan group

SUMMARY:
Hypertension is the most common complication in patients with diabetes nephropathy. Strengthening blood pressure and blood sugar control is the basic treatment for patients with diabetes nephropathy. Angiotensin receptor blocker (ARB) and angiotensin-converting enzyme inhibitor (ACEI) are the first line drugs recommended in domestic and international guidelines for diabetes patients to control hypertension. As a new ARB drug, azilsartan has been found to have better antihypertensive effect than other ARB drugs. However, due to the limited sample size and study time, azilsartan has no significant advantage over other ARB drugs in terms of renal protection effect, and has not been systematically studied in diabetes nephropathy population. This study is intended to evaluate the effect of azilsartan on proteinuria and blood pressure improvement in patients with diabetes nephropathy and hypertension through clinical randomized controlled study, so as to accumulate evidence-based evidence of azilsartan in the comprehensive management of heart and kidney protection in this group of people, and promote the development of comprehensive treatment for patients with metabolic disease and renal injury combined with hypertension. This study will compare the advantages and disadvantages of azilsartan and classical ARB drug losartan potassium in terms of proteinuria, blood pressure control and renal function protection in patients with diabetes nephropathy and hypertension; We propose that the main indicator is the change of urinary albumin/creatinine ratio relative to the baseline, and the secondary indicator is the change of 24-hour urinary protein relative to the baseline; Change of blood pressure relative to baseline; Renal function, electrolyte and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 70;
* Type 2 diabetes diagnosed according to American Diabetes Association guidelines has stable blood sugar control, and glycosylated hemoglobin is less than 7.5%;
* The patient's blood pressure Systemic Blood Pressure (SBP) >140 or Diastolic Blood Pressure (DBP) >90 mmHg, has not taken antihypertensive drugs or is taking non-ARB/ACEI antihypertensive drugs;
* Urine albumin/creatinine ratio>300mg/g.

Exclusion Criteria:

* Type 1 diabetes;
* The patient is considered as non-essential hypertension, such as hypertension caused by renal hypertension or endocrine disease;
* Contraindications of ARB drugs, such as pregnancy status, bilateral renal artery stenosis, allergy to ARB drugs and their excipients;
* It is expected that dialysis treatment will be carried out within 6 months;
* Patients with malignant tumors;
* Patients with mental illness;
* The researcher believes that others are not suitable for this study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
proteinuria | up to 16 weeks
  urinary protein

SECONDARY OUTCOMES:
24 hour urine protein | up to 16 weeks
  24 hour total protein
blood pressure | up to 16 weeks
  bp
kidney function | up to 16 weeks
  creatine, Blood Urine Nitrogen
urinary albumin/ creatine | up to 16 weeks
  urinary albumin/ creatine

CONTACTS AND LOCATIONS:
Overall Officials: Zhida Chen, Principal Investigator — The second afiliated hospital of zhejiang university, school of medicine
Locations (1):
- the Second Afficiated Hospital, Zhejiang University, School of Medicine, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786